CLINICAL TRIAL: NCT06629389
Title: Randomized, Double-blind, Placebo-controlled, Phase II Clinical Trial to Evaluate Safety and Tolerability of Cannabidiol (Kanbis®) for the Treatment of Parkinson's Disease Symptoms
Brief Title: Clinical Trial with Cannabidiol (Kanbis®) for Parkinson Disease Symptoms
Acronym: CBD-EP-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-EP-2
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; Cannabidiol; oil; cannabis
MeSH Terms: conditions — Parkinson Disease; Marijuana Abuse | interventions — Cannabidiol; nabiximols

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group CBD 100 (Active Comparator): The following dose regime for the 4 treatment arms will be used
  Interventions: Drug: Cannabidiol 100 mg/ml
- Group CBD 300 (Active Comparator): The following dose regime for the 4 treatment arms will be used
  Interventions: Drug: cannabidiol 300 mg/ml
- Group CBD 400 (Active Comparator): The following dose regime for the 4 treatment arms will be used
  Interventions: Drug: Cannabidiol 100 mg/ml; Drug: Cannabidiol 400 mg/ml
- Group Placebo (Placebo Comparator): The following dose regime for the 4 treatment arms will be used
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol 100 mg/ml — The following dose regime for the 4 treatment arms will be used:
  DOSE TITRATION PERIOD:
  First 5 days: 0.3 mL/day (1 dose) Subsequent 5 days: 0.6 mL/day (2 doses of 0.3 mL/dose) Subsequent 5 days: 0.8 mL/day (2 doses of 0.4 mL/dose) Last 5 days: 1 mL/day (2 doses of 0.4 mL/dose) PERIOD OF ACTIVE TREATMENT Continue with the last dose set by the titration schedule (for 12 weeks). PERIOD OF TREATMENT INTERRUPTION Medication is gradually discontinued every 7 days until complete termination. The first 7 days dose will be reduced to 0.5 mL/day; on subsequent 7 days, dose will be reduced to 0.3 mL/day. If a patient has reached a maximum tolerated dose, dose reduction will be made at the discretion of the investigator.
  Other Names: CBD; Cannabis
  Arms: Group CBD 100; Group CBD 400
Drug: cannabidiol 300 mg/ml — The following dose regime for the 4 treatment arms will be used:
  DOSE TITRATION PERIOD:
  First 5 days: 0.3 mL/day (1 dose) Subsequent 5 days: 0.6 mL/day (2 doses of 0.3 mL/dose) Subsequent 5 days: 0.8 mL/day (2 doses of 0.4 mL/dose) Last 5 days: 1 mL/day (2 doses of 0.4 mL/dose) PERIOD OF ACTIVE TREATMENT Continue with the last dose set by the titration schedule (for 12 weeks). PERIOD OF TREATMENT INTERRUPTION Medication is gradually discontinued every 7 days until complete termination. The first 7 days dose will be reduced to 0.5 mL/day; on subsequent 7 days, dose will be reduced to 0.3 mL/day. If a patient has reached a maximum tolerated dose, dose reduction will be made at the discretion of the investigator.
  Arms: Group CBD 300
Drug: Cannabidiol 400 mg/ml — The following dose regime for the 4 treatment arms will be used:
  DOSE TITRATION PERIOD:
  First 5 days: 0.3 mL/day (1 dose) Subsequent 5 days: 0.6 mL/day (2 doses of 0.3 mL/dose) Subsequent 5 days: 0.8 mL/day (2 doses of 0.4 mL/dose) Last 5 days: 1 mL/day (2 doses of 0.4 mL/dose) PERIOD OF ACTIVE TREATMENT Continue with the last dose set by the titration schedule (for 12 weeks). PERIOD OF TREATMENT INTERRUPTION Medication is gradually discontinued every 7 days until complete termination. The first 7 days dose will be reduced to 0.5 mL/day; on subsequent 7 days, dose will be reduced to 0.3 mL/day. If a patient has reached a maximum tolerated dose, dose reduction will be made at the discretion of the investigator.
  Arms: Group CBD 400
Drug: Placebo — The following dose regime for the 4 treatment arms will be used:
  DOSE TITRATION PERIOD:
  First 5 days: 0.3 mL/day (1 dose) Subsequent 5 days: 0.6 mL/day (2 doses of 0.3 mL/dose) Subsequent 5 days: 0.8 mL/day (2 doses of 0.4 mL/dose) Last 5 days: 1 mL/day (2 doses of 0.4 mL/dose) PERIOD OF ACTIVE TREATMENT Continue with the last dose set by the titration schedule (for 12 weeks). PERIOD OF TREATMENT INTERRUPTION Medication is gradually discontinued every 7 days until complete termination. The first 7 days dose will be reduced to 0.5 mL/day; on subsequent 7 days, dose will be reduced to 0.3 mL/day. If a patient has reached a maximum tolerated dose, dose reduction will be made at the discretion of the investigator.
  Arms: Group Placebo

SUMMARY:
Parkinson disease (PD) is a chronic, progressive neurodegenerative disorder characterized by clinical motor and non-motor symptoms. Knowing the potential benefits has led to the use of cannabis as an alternative therapy.

DETAILED DESCRIPTION:
To evaluate safety and tolerability of CBD-based drug product at different doses

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 40 and 80 years old.
2. Participants diagnosed with PD according to Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease (72), and to the Brain Bank Criteria for Parkinson's disease, with mild to moderate disease as measured by the modified Hoehn and Yahr scale. (Both clinical criteria are included since many of the study participants were diagnosed with previous criteria and others with current criteria, both of which are very similar and do not change or raise any doubt about the diagnosis of the disease).
3. Participants who have not changed their anti-Parkinson's drugs (or dose) at least one month prior to study entry.
4. Acceptance by the participant by signing the ICF.
5. Subjects capable of giving consent to participate in the study

Exclusion Criteria:

1. Evidence of dementia, Mini-Mental State Exam score less than 24 or with previous diagnosis by cognitive assessment .
2. Severe psychiatric pathology: severe depression, treatment-refractory psychosis. Evaluation by psychiatrist who confirms the pathology. History of hospitalization in a psychiatric center or mental health center is an exclusion criterion regardless of the time spent since hospitalization or the reason for which the patient was hospitalized.
3. Known or suspected allergy to cannabinoids or inactive ingredients used in the formulation of the study drug.
4. History of drug or alcohol dependence.
5. Use of dopamine blockers within 180 days prior to study entry.
6. Use of amphetamine inhibitors, cocaine and MAO-A inhibitors within 90 days prior to study entry.
7. Patients who have received within 90 days prior to study entry the following drugs due to drug interactions: valproic acid, felbamate, niacin (nicotinic acid) at doses ≥2000mg/day or nicotinamide (nicotinic acid amide or nicotinamide) at doses ≥3000mg/day, isoniazid, ketoconazole and/or clobazam.
8. Unstable medical condition detected by the following laboratory alterations: Hemoglobin<10g/dL, Leukocytes<4000 u/ml, Neutrophils<1500 u/ml, Lymphocytes<500u/ml, Platelets<100000 u/ml, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)> 3 times the upper limit of normal.
9. Moderate-severe liver disease. (Child Pugh B-C)
10. Pregnant or breastfeeding.
11. Women of reproductive age who do not agree to use at least one contraceptive method of proven efficacy (diaphragm or partner using condom, oral or implanted hormonal contraceptive; intrauterine device, stable partner with vasectomy), until at least four weeks after completion of study treatment. Pregnancy blood test will be performed before starting the study.
12. Participants who have had a surgical procedure for PD, either deep brain stimulation or surgery for lesion.
13. Patients de novo or with recent diagnosis of PD (less than 5 years).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with advers events related to treatment acording to CTCAE v5.0 | up to 21 weeks
  Frequency of adverse events by a global comparison of all dose or placebo groups Range: 1 to 5 Higher values represent a worse disease state

SECONDARY OUTCOMES:
Changes in differents motors scales in Parkinson desease | up to 15 weeks
  changes in the Unified Parkinson's Disease Rating Scale scale (MDS-UPDRS) part I (mental section), part II (daily activities), part III, (motor section), and part IV (treatment complications).
  Overall range (Part I+II+III+IV): 0 to 260 Higher values represent a worse disease state
Changes in the off periods in Parkinson desease | up to 15 weeks
  • variations in the off periods using the patient's personal diary
Changes in the patients Clinical Global Impression in Parkinson desease | up to 21 weeks
  • changes in the patients Clinical Global Impression as measured by the Clinical Global Impression-Severity Scale (CGI-S).
  Range: 0 to 7 Higher values represent a worse disease state
Changes in the quality-of-life in Parkinson desease | up to 15 weeks
  • changes in the quality-of-life scale with the Parkinson's Disease Questionnaire (PDQ39).
  Range: 0 to 100 Higher values represent a worse disease state
Changes in differents no motors symproms in Parkinson desease | up to 15 weeks
  • changes in non-motor symptoms by means of Non-Motor Symptom Scale (NMSS) and Non-Motor Symptoms Questionnaire (NMSQ).
Changes in depression in Parkinson desease | up to 15 weeks
  • changes in depression with the Beck Depression Inventory Scale (BDI-II). Overall range: 0 to 63. Higher values represent a worse disease state
Changes in sleep in Parkinson disease | up to 15 weeks
  • changes in the sleep scale for Parkinson Desease with Epworth Scale. Overall range: 0 to 24. Higher values represent a worse disease state
Changes in Cognitive Assessment in Parkinson desease | up to 15 weeks
  To assess the Montreal Cognitive Assessment (MoCA) scale Maximum score 30 Score greater than 26 is considered normal
Changes in apathy in Parkinson desease | up to 15 weeks
  • changes in apathy measured by the Apathy Evaluation Scale (AES). Total score ranges: 18 to 72 Higher scores indicating more apathy
Changes in pain in Parkinson desease | up to 15 weeks
  • DP pain-related changes measured by the King's Parkinson's Disease Pain Scale (KPSS).
  Range: 0 to 168 Higher values represent a worse disease state

CONTACTS AND LOCATIONS:
Overall Officials: Marina Sanchez Abraham, Neurologa, Principal Investigator — Hospital Español de Mendoza
Locations (1):
- Hospital Español de Mendoza, Mendoza, Mendoza Province, Argentina

IPD SHARING:
Plan to Share IPD: No